CLINICAL TRIAL: NCT01114269
Title: PRE-DETERMINE: Biologic Markers and MRI SCD Cohort Study
Brief Title: PRE-DETERMINE Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Abbott Medical Devices (Industry); Northwestern University (Other); Quintiles, Inc. (Industry); Roche Diagnostic Ltd. (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Christine M. Albert, MD, MPH, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2007P000840; R01HL091069 (NIH); R01HL165840 (NIH)
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease; Left Ventricular Dysfunction; Sudden Cardiac Death
Keywords: Coronary Artery Disease; Sudden Cardiac Death; Myocardial Infarction; Percutaneous Coronary Intervention; Implantable Cardiac Defibrillator
MeSH Terms: conditions — Coronary Artery Disease; Ventricular Dysfunction, Left; Death, Sudden, Cardiac; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, buffy coat, and red blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, multi-center cohort study of patients with a history of coronary artery disease (CAD) and documentation of either a prior myocardial infarction (MI) or mild to moderate left ventricular dysfunction (LVEF 35-50%). The primary objective of this study is to determine whether biologic markers and ECGs can be utilized to advance SCD risk prediction in patients with CHD and LVEF>30-35%. The overarching goal of the study is to identify a series of markers that alone or in combination specifically predict risk of arrhythmic death as compared to other causes of mortality among this at risk population of coronary heart disease (CHD) patients with preserved left ventricular ejection fraction (LVEF> 30-35%). If biologic or ECG markers are identified that can specifically predict risk of ventricular arrhythmias, then these markers may serve as relatively inexpensive methods to identify those at risk. The public health impact of identifying markers could be quite substantial, leading to more efficient utilization of ICDs and advances in our understanding of mechanisms underlying SCD.

DETAILED DESCRIPTION:
The PRE-DETERMINE Study is a prospective, multi-center study of patients with a history of coronary artery disease (CAD) and documentation of either a prior myocardial infarction (MI) or mild to moderate left ventricular dysfunction (LVEF 35-50%). Patients were enrolled at 135 sites where information on baseline demographics, clinical characteristics, pertinent past medical history, lifestyle habits, cardiac test results, and medications were collected via electronic data capture. Electrocardiograms along with a blood sample was also collected at baseline, sent to central laboratories, and stored for future analyses. Contrast-enhanced magnetic resonance imaging (CE-MRI) scans were collected on a subset of patients and analyzed. Enrollment closed in November 2013 and patients are now being followed centrally by the Clinical Coordinating Center via mail/phone to document interim non-fatal arrhythmic events and cause-specific mortality. Questionnaires that inquire about intervening ICD implantations, ICD therapies, cardiac arrest, and other pertinent cardiovascular endpoints are mailed to participants every six months, and follow-up telephone calls are made to non-responders. Study endpoints are being confirmed through review of medical records, interviews with next-of-kin, and autopsy reports, if available.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of Coronary Artery Disease (CAD) a or documented prior Myocardial Infarction.
2. LVEF >35% by any current standard evaluation technique (e.g.,) echocardiogram, MUGA, angiography). 2.1. Patients who have an LVEF between 30-35% and NYHA Class I heart failure who do not have history of ventricular tachyarrhythmias,or inducible ventricular tachycardia during electrophysiological (EP) testing can be enrolled.
3. If documented prior MI is not present, evidence of mild-moderate systolic Left Ventricular Dysfunction with an EF >35- ≤50% as measured by any current standard screening technique (e.g.,echocardiogram, MUGA, angiography) must be present.
4. Patients aged 18 years or above

   1. CAD will be defined as evidence of one of the following two (2) criteria:

      * Significant stenosis of a major epicardial vessel (>50% proximal or 70% distal) by coronary angiography
      * Prior revascularization (percutaneous coronary intervention or coronary artery bypass surgery)
   2. MI can be documented in the following ways:

      * From the MI hospitalization: Detection of a rise and fall of cardiac biomarkers > 99th percentile of lab (e.g., CPK elevation or Troponin at least > two times the upper limit of normal) together with myocardial ischemia with at least one of the following:

        * Symptoms of Ischemia
        * ECG changes indicative of new ischemia (new ST-T changes or new LBBB)
        * Development of pathological Q waves
        * Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality
      * If no report from the MI hospitalization is available, prior MI can be met by either of the following:

        * Development of pathological Q waves
        * Imaging evidence of a region of loss of viable myocardium that is thinned and fails to contract, in the absence of a non-ischaemic cause

Exclusion Criteria:

1. History of cardiac arrest or spontaneous or inducible sustained VT (15 beats or more at a rate of 120 BPM or greater - the occurrence of cardiac arrest or spontaneous VT in the setting of an acute MI is not considered an exclusion).
2. Unexplained syncope
3. Current or planned implantable cardiac defibrillator (ICD)
4. Any condition other than cardiac disease that, in the investigator's judgment, would seriously limit life expectancy (poor survival)
5. Metastatic cancer
6. Marked valvular heart disease requiring surgical intervention
7. Current or planned cardiac, renal or liver transplant
8. Current alcohol or drug abuse
9. Unwilling or unable to provide informed consent
10. LVEF <35% with Class II-IV CHF or LVEF <30%
11. Participation in a clinical trial where the active treatment arm is testing an agent and/or intervention with known antiarrhythmic properties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants have been recruited throughout multicenter sites participating in the PRE-DETERMINE Cohort Study. Patients with a history of coronary artery disease and documentation of either a prior myocardial infarction (MI) or mild to moderate left ventricular dysfunction (LVEF 35-50%) have been enrolled. The clinical study staff at each site, which was either a research nurse, fellow, or physician approached eligible patients to discuss their potential participation.
Sampling Method: Probability Sample
Enrollment: 5764 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Sudden and/or arrhythmic cardiac death or resuscitated ventricular fibrillation. | Median follow-up estimated to be 10.7 years
  A definite sudden cardiac death (SCD) is defined as a death or fatal cardiac arrest occurring within 1 hour of symptom onset or the presence of autopsy consistent with SCD (e.g. acute coronary thrombosis). Probable SCD is defined as an unwitnessed death or death during sleep where the participant was observed to be symptom-free within the preceding 24 hours. Arrhythmic death is defined as the abrupt spontaneous collapse of circulation without antecedent circulatory or neurologic impairment. Deaths classified as non-arrhythmic are not included in the primary endpoint regardless of timing. Resuscitated ventricular fibrillation is defined as out-of-hospital cardiac arrests with documented VF and/or use of external electrical defibrillation for resuscitation.

SECONDARY OUTCOMES:
ICD Shock | Median follow-up estimated to be 10.7 years
  ICD therapies for ventricular arrhythmias over 200 BPMs will be added to the endpoint.
ICD Implantation | Median follow-up estimated to be 10.7 years
Total Cardiac Mortality | Median follow-up estimated to be 10.7 years
Total Mortality | Median follow-up estimated to be 10.7 years
Non-Sudden or Arrhythmic Causes of Mortality | Median follow-up estimated to be 10.7 years
  Competing causes of mortality in competing risk analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Albert, M.D., M.P.H., Principal Investigator — Brigham and Women's Hospital
Locations (90):
- United States (86):
  - Alaska Heart Institute, Anchorage, Alaska
  - Phoenix Heart, PLLC, Glendale, Arizona
  - Cardiovascular Consultants, Phoenix, Arizona
  - Beaver Medical Group/Clinical Care Research, Banning, California
  - Memorial Health System, Colorado Springs, Colorado
  - Colorado Heart and Vascular, Denver, Colorado
  - Bay Area Cardiology Associates, P.A., Brandon, Florida
  - University of Florida - Gainsville, Gainesville, Florida
  - Reliable Clinical Research, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital, Orlando, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Palm Beach Gardens Research Center, Palm Beach Gardens, Florida
  - Velella Research, Sarasota, Florida
  - Tallahassee Research Institute, Inc., Tallahassee, Florida
  - Cardiology Associates of Palm Beach - West Palm Beach, West Palm Beach, Florida
  - Georgia Heart Specialist, Covington, Georgia
  - Northeast Georgia Heart Center, P.C., Gainesville, Georgia
  - University of Chicago, Chicago, Illinois
  - Advocate Medical Group, Chicago, Illinois
  - Advocate Medical Group - Heart and Vascular of IL, Chicago, Illinois
  - Consultants in Cardiovascular Medicine, Melrose Park, Illinois
  - Community Heart and Vascular, Anderson, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - The University of Kansas, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Leonard J. Chabert Medical Center, Houma, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Maine Research Associates - Lewiston, Lewiston, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Primary Care Cardiology Research, Ayer, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - NECCR Internal Medicine and Cardiology Associates, LLC, Fall River, Massachusetts
  - Hawthorn Medical Associates, North Dartmouth, Massachusetts
  - Baystate Cardiology, Springfield, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Oakwood Hospital & Medical Center, Dearborn, Michigan
  - McLaren Medical Center - Macomb, Mount Clemens, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - Glacier View Cardiology, Kalispell, Montana
  - The Cardiac Center of Creighton University, Omaha, Nebraska
  - Advanced Heartcare, LLC, Bridgewater, New Jersey
  - St. Joseph Regional Medical Center, Paterson, New Jersey
  - New Mexico VA Healthcare Systems, Albuquerque, New Mexico
  - Albany Associates Cardiology, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Buffalo General Hospital/Kaleida Health, Buffalo, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Mid-Valley Cardiology, Kingston, New York
  - Winthrop-University Hospital, Mineola, New York
  - Gotham Cardiovascular, New York, New York
  - Columbia University Health Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - St. Elizabeth Medical Center - Hotvedt, Utica, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Eastern Carolina Cardiovascular, Elizabeth City, North Carolina
  - Northstate Clinical Research, Lenoir, North Carolina
  - Pinehurst Medical Clinic, Inc., Pinehurst, North Carolina
  - Sanford Cardiology, Sanford, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - Northeast Ohio Cardiovascular Specialists, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - North Ohio Research, Ltd., Elyria, Ohio
  - Mercy Medical Associates, Fairfield, Ohio
  - Northwest Ohio Cardiology Consultants/The Toledo Hospital, Toledo, Ohio
  - Oklahoma City VA Medical Center Veterans Research and Education Foundation, Oklahoma City, Oklahoma
  - Oklahoma Foundation for Cardiovascular Research, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - St. Luke's Bethlehem, Bethlehem, Pennsylvania
  - Doylestown Cardiology Associates, Doylestown, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - VA Medical Center - Charleston, Charleston, South Carolina
  - Carolina Cardiology Associates, Rock Hill, South Carolina
  - Black Hills Cardiovascular Research, Rapid City, South Dakota
  - Cardiovasular Research of Knoxville, Knoxville, Tennessee
  - Memphis VA Medical Center, Memphis, Tennessee
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Non-Invasive Cardiovascular PA, Houston, Texas
  - Providence Health Center, Waco, Texas
  - Intermountain Medical Center, Murray, Utah
  - Cardiovascular Associates Virginia Beach, Virginia Beach, Virginia
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Mississauga Clinical Research Centre, Mississauga, Ontario
- Transcatheter Medical, Inc. Centro Cardiovascular de Caguas y del Caribe, Rio Piedras, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krieglstein GK, Schrems W. [Stereospecificity of beta-blocker effects on the glaucomatous eye]. Fortschr Ophthalmol. 1984;81(2):127-9. No abstract available. German. PMID 6145665
- [Result] Friedlander MH, Werblin TP, Kaufman HE, Granet NS. Clinical results of keratophakia and keratomileusis. Ophthalmology. 1981 Aug;88(8):716-20. doi: 10.1016/s0161-6420(81)34957-4. PMID 7033860
- [Result] Weisgraber KH, Rall SC Jr, Mahley RW. Human E apoprotein heterogeneity. Cysteine-arginine interchanges in the amino acid sequence of the apo-E isoforms. J Biol Chem. 1981 Sep 10;256(17):9077-83. No abstract available. PMID 7263700
- [Result] Chao FC, Tullis JL, Alper CA, Glynn RJ, Silbert JE. Alteration in plasma proteins and platelet functions with aging and cigarette smoking in healthy men. Thromb Haemost. 1982 Jun 28;47(3):259-64. PMID 6981228
- [Result] Sandhu RK, Dron JS, Liu Y, Moorthy MV, Chatterjee NA, Ellinor PT, Chasman DI, Cook NR, Khera AV, Albert CM. Polygenic Risk Score Predicts Sudden Death in Patients With Coronary Disease and Preserved Systolic Function. J Am Coll Cardiol. 2022 Aug 30;80(9):873-883. doi: 10.1016/j.jacc.2022.05.049. PMID 36007985
- [Result] Peek N, Hindricks G, Akbarov A, Tijssen JGP, Jenkins DA, Kapacee Z, Parkes LM, van der Geest RJ, Longato E, Sprague D, Taleb Y, Ong M, Miller CA, Shamloo AS, Albert C, Barthel P, Boveda S, Braunschweig F, Johansen JB, Cook N, de Chillou C, Elders P, Faxen J, Friede T, Fusini L, Gale CP, Jarkovsky J, Jouven X, Junttila J, Kautzner J, Kiviniemi A, Kutyifa V, Leclercq C, Lee DC, Leigh J, Lenarczyk R, Leyva F, Maeng M, Manca A, Marijon E, Marschall U, Merino JL, Mont L, Nielsen JC, Olsen T, Pester J, Pontone G, Roca I, Schmidt G, Schwartz PJ, Sticherling C, Suleiman M, Taborsky M, Tan HL, Tfelt-Hansen J, Thiele H, Tomaselli GF, Verstraelen T, Vinayagamoorthy M, Olesen KKW, Wilde A, Willems R, Wu KC, Zabel M, Martin GP, Dagres N. Sudden cardiac death after myocardial infarction: individual participant data from pooled cohorts. Eur Heart J. 2024 Nov 14;45(43):4616-4626. doi: 10.1093/eurheartj/ehae326. PMID 39378245
- [Result] Panicker GK, Narula DD, Albert CM, Lee DC, Kothari S, Goldberger JJ, Cook N, Schaechter A, Kim E, Moorthy MV, Pester J, Chatterjee NA, Kadish AH, Karnad DR. Validation of electrocardiographic criteria for identifying left ventricular dysfunction in patients with previous myocardial infarction. Ann Noninvasive Electrocardiol. 2021 Mar;26(2):e12812. doi: 10.1111/anec.12812. Epub 2020 Oct 30. PMID 33124739
- [Result] Venkateswaran RV, Moorthy MV, Chatterjee NA, Pester J, Kadish AH, Lee DC, Cook NR, Albert CM. Diabetes and Risk of Sudden Death in Coronary Artery Disease Patients Without Severe Systolic Dysfunction. JACC Clin Electrophysiol. 2021 Dec;7(12):1604-1614. doi: 10.1016/j.jacep.2021.05.014. Epub 2021 Jul 28. PMID 34332876
- [Derived] Chatterjee NA, Tikkanen JT, Panicker GK, Narula D, Lee DC, Kentta T, Junttila JM, Cook NR, Kadish A, Goldberger JJ, Huikuri HV, Albert CM; PREDETERMINE Investigators. Simple electrocardiographic measures improve sudden arrhythmic death prediction in coronary disease. Eur Heart J. 2020 Jun 1;41(21):1988-1999. doi: 10.1093/eurheartj/ehaa177. PMID 32259257
- [Derived] Adabag S, Patton KK, Buxton AE, Rector TS, Ensrud KE, Vakil K, Levy WC, Poole JE. Association of Implantable Cardioverter Defibrillators With Survival in Patients With and Without Improved Ejection Fraction: Secondary Analysis of the Sudden Cardiac Death in Heart Failure Trial. JAMA Cardiol. 2017 Jul 1;2(7):767-774. doi: 10.1001/jamacardio.2017.1413. PMID 28724134
- See also: Cardiac Arrest — http://www.nlm.nih.gov/medlineplus/cardiacarrest.html
- See also: Coronary Artery Disease — http://www.nlm.nih.gov/medlineplus/coronaryarterydisease.html
- See also: Pacemakers and Implantable Defibrillators — http://www.nlm.nih.gov/medlineplus/pacemakersandimplantabledefibrillators.html
- See also: U.S. FDA Resources — http://clinicaltrials.gov/ct2/info/fdalinks
- See also: Heart Disease — http://www.nlm.nih.gov/medlineplus/heartdiseases.html
- See also: PRE-DETERMINE Study Website — https://www.pre-determinestudy.org